CLINICAL TRIAL: NCT00035529
Title: A Phase II,Randomized, Double-Blind, Placebo Controlled Study to Evaluate the Preliminary Efficacy, Pharmacokinetics and Immunogenicity of BMS-188667 Administered to Subjects With Relapsing-Remitting Multiple Sclerosis
Brief Title: A Study to Evaluate the Preliminary Efficacy Pharmacokinetics and Immunogenicity of BMS-188667 Administered to Subjects With Relapsing-remitting Multiple Sclerosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM101-200
Record Dates: First submitted 2002-05-03; First posted 2002-05-06 (Estimated); Last update posted 2010-12-06 (Estimated); Status verified 2010-12

CONDITIONS: Multiple Sclerosis
Keywords: MS
MeSH Terms: conditions — Multiple Sclerosis | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Other)
  Interventions: Drug: Placebo
- 2 (Active Comparator)
  Interventions: Drug: BMS 188667 (Abatacept)
- 3 (Active Comparator)
  Interventions: Drug: BMS 188667 (Abatacept)

INTERVENTIONS:
Drug: Placebo — Solution, i.v infusion, 0 mg, Days 1 & 15 then monthly, 10 months.
  Arms: 1
Drug: BMS 188667 (Abatacept) — Vial, i.v infusion, 2mg/kg, Days 1 & 15 then monthly, 10 months.
  Other Names: Orencia
  Arms: 2
Drug: BMS 188667 (Abatacept) — Vial, i.v infusion, 10 mg/kg, Days 1 & 15 then monthly, 10 months.
  Other Names: Orencia
  Arms: 3

SUMMARY:
The purpose of this study is to determine whether BMS-188667 will decrease multiple sclerosis disease activity on MRI examinations, as well as decrease the rate of clinical MS exacerbations, compared to placebo

ELIGIBILITY:
Inclusion

* relapsing-remitting MS
* at least 1 exacerbation in preceding 2 years
* at least 1 MRI lesion
* stable for 2 months prior to dosing

Exclusion

* progressive MS
* currently treated with an immunomodulatory therapy
* previously treated with an approved MS drug where treatment was discontinued for lack of efficacy
* active bacterial or viral infections

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2001-11; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Preliminary efficacy- Reduction in cumulative nr of new or recurrent Gd-enhancing lesions.

SECONDARY OUTCOMES:
Preliminary efficacy: 1) Decrease in annualized relapse rate and 2) Reduction in cumulative nr of new or enlarging T2-weighted MRI lesions.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Local Institution, New Haven, Connecticut
  - Local Institution, Louisville, Kentucky
  - Local Institution, Worcester, Massachusetts
  - Local Institution, Newark, New Jersey
  - Local Institution, New York, New York
  - Local Institution, Charlotte, North Carolina
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Dallas, Texas
  - Local Institution, Burlington, Vermont
  - Local Institution, Madison, Wisconsin